CLINICAL TRIAL: NCT04846751
Title: Exercise Type That Faster Reduces Postprandial Glycemia.
Acronym: GLYEXER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Ricardo Mora, Director of the Exercise Lab at Toledo, University of Castilla-La Mancha
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PID2020-116159RB-I00
Record Dates: First submitted 2021-04-11; First posted 2021-04-15 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Glucose, High Blood; Exercise-Induced Hyperinsulinism
MeSH Terms: conditions — Hyperinsulinemic hypoglycemia, familial, 7

STUDY DESIGN:
Intervention Model Description: Study composed of 4 trials, full-crossover, administered in a randomized order with the inclusion of a control trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AEROBIC EXERCISE (Active Comparator): 50 min of aerobic exercise by pedaling a cycleergometer at 60% of VO2max
  Interventions: Behavioral: TYPE OF EXERCISE (OR REST)
- PLACEBO REST (Placebo Comparator): No exercise, resting during 50 min.
  Interventions: Behavioral: TYPE OF EXERCISE (OR REST)

INTERVENTIONS:
Behavioral: TYPE OF EXERCISE (OR REST) — continous exercise in normal temperature, continous exercise in hot environment, intervallic exercise in normal temperature.

SUMMARY:
It is well established that a bout of 50 min of continuous moderate intensity exercise, improves insulin sensitivity up to 48 hours after the bout. However, it is less well known, what is the exercise type more efficient to buffer the elevations in blood glucose elicited by carbohydrate ingestion. The purpose of this study is to elucidate if intervalic exercise is superior to continous on improving postprandial glycemic control.

DETAILED DESCRIPTION:
Carbohydrate oxidation, glucose and insulin blood concentrations, isotopically measured rate of appearance of endogenous and exogenous glucose will be measured in 4 ocassions.

Participants will undergo in a cross-over randomized fashion the following trials:

1. Exercise pedalling during 50 min at 60% of their VO2max followed by an oral glucose tolerance test (OGTT).
2. Exercise pedalling during 50 min in a hot environment (33ºC) at 60% of their VO2max followed by an oral glucose tolerance test (OGTT).
3. Exercise pedalling during 50 min using intervalic bouts averaging 60% of VO2max followed by an oral glucose tolerance test (OGTT).
4. No exercise, followed by an oral glucose tolerance test (OGTT).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be capable and willing to provide consent, understand, instructions and protocols.
* Minimal fitness level to be able to complete 50 min of continous exercise at a moderate intensity.

Exclusion Criteria:

* Smokers
* Pregnancy
* Any non-controlled medical condition which could influence results or could be worsened by exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Blood glucose concentration | 16 weeks
  Incremental area under the curve during the 120 min of the oral glucose tolerance test
Blood insulin concentration | 16 weeks
  Incremental area under the curve during the 120 min of the oral glucose tolerance test

SECONDARY OUTCOMES:
Carbohydrate oxidation | 16 weeks
  Measured using indirect calorimetry
Turnover rate of endogenous and exogenous glucose | 16 weeks
  Measured using isotopic tracers.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Mora-Rodriguez, PhD, Principal Investigator — University of Castilla-La Mancha
Locations (1):
- University of Castilla-La Mancha (Exercise Physiology Lab), Toledo, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon reasonable request.